CLINICAL TRIAL: NCT06098378
Title: Retrospective Study of Patients With Thrombotic Microangiopathy Associated With Mitomycin C, Treated or Not With Eculizumab: Clinical Characteristics and and Outcome of These Patients
Brief Title: Study of Patients With Thrombotic Microangiopathy Associated With Mitomycin C, Treated or Not With Eculizumab
Acronym: m-TMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8957
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Thrombotic Microangiopathies
Keywords: Thrombotic Microangiopathies; Mitomycin C; Mitomycin-C-induced TMA; m-TMA; Eculizumab; Hemolytic uremic syndrome
MeSH Terms: conditions — Thrombotic Microangiopathies; Hemolytic-Uremic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thrombotic microangiopathies (TMA) are defined as a triad combining mechanical hemolytic anemia, peripheral thrombocytopenia and ischemic organ damage.

Mitomycin C is an alkylating agent used as chemotherapy in adenocarcinomas of the breast, lung, pancreas, rectum and anal carcinoma. Mitomycin-C-induced TMA (m-TMA) is a potentially serious complication of chemotherapy: its estimated incidence ranges from 4 to 15% and its mortality exceeds 70%, with an estimated median survival of 2 months. This can also be responsible for kidney failure, sometimes requiring hemodialysis. The time to onset of m-TMA varies from one week to 15 months after the last infusion and is believed to depend on the cumulative dose of mitomycin C.

Eculizumab is a monoclonal antibody that binds to complement protein C5, blocking activation of the terminal complement pathway and formation of the membrane attack complex. This therapy has significantly changed the prognosis of patients with atypical hemolytic uremic syndrome (HUS), a disease in which complement activation plays a central role in TMA. Recently, a retrospective study suggested efficacy of eculizumab in TMA induced by gemcitabine, another chemotherapy, with normalization of platelets and LDH in 83% of patients, and partial or complete renal recovery in 67% and 17% of patients. These results provided arguments in favor of a potential benefit of complement-targeted therapies in TMA induced by certain chemotherapies. However, data on eculizumab in m-TMA remain extremely limited to date.

The objective of this study is to describe the clinical, biological and histological presentation of patients with m-TMA and their evolution after treatment with or without eculizumab.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>=18 years)
* Having received treatment with mitomycin C (regardless of the method of administration and indication) between 01/01/1990 and 12/31/2023
* and having developed a picture of thrombotic microangiopathy attributed to mitomycin C:

  * biological: defined as: thrombocytopenia <150G/L and mechanical hemolytic anemia (at least 3 out of 4 criteria: hemoglobin < 12g/dL, presence of schistocytes in blood smear, LDH > 1N, collapsed haptoglobin (< lower limit of the limit of laboratory normal)
  * or renal: pathological diagnosis of thrombotic microangiopathy on renal biopsy
* having received or not treatment for the episode of microangiopathy, including or not complement inhibitors (Eculizumab).
* Subject not opposing, after information, the reuse of their data for the purposes of this research

Exclusion Criteria:

* Subject having expressed opposition to participating in the study
* Test for positive Shiga toxin
* ADAMST13 activity <10%
* Thrombotic microangiopathy attributed to metastatic cancer (infiltration of bone marrow or circulating erythroblasts)
* Impossibility of providing the subject with informed information (difficulties in understanding the subject, etc.)
* Subject under judicial protection
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients (>=18 years) having developed a picture of thrombotic microangiopathy attributed to mitomycin C between 01/01/1990 and 12/31/2023
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06-07 (Estimated)

PRIMARY OUTCOMES:
Overall and renal survival after the m-TMA episode | Files analysed retrospectively from January 01, 1990 to December 31, 2023 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Néphrologie, Dialyse et Transplantation - CHU de Strasbourg - France, Strasbourg, France